CLINICAL TRIAL: NCT01801345
Title: The Effect of Fatigue on the Clinical Performance of Experienced Physicians: A Simulation Study
Brief Title: The Effect of Fatigue on the Clinical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EH12-048
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Fatigue
Keywords: Human Performance; Clinical Performance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rested (Other): Subjects will perform the scenario, once during a normal workday (rested)
  Interventions: Other: Rested
- Fatigued (Active Comparator): Subjects will perform the scenario after working a 12-24 hour overnight shift (fatigued).
  Interventions: Other: Fatigued

INTERVENTIONS:
Other: Fatigued
  Arms: Fatigued
Other: Rested
  Arms: Rested

SUMMARY:
The primary aim of this randomized controlled trial is to examine the effect of fatigue on clinical performance in a simulated obstetric emergency. This scenario was chosen because it is a common clinical situation faced by anesthesia providers on call and therefore likely to occur when a provider is fatigued. Secondary outcomes will include the evaluation of other factors that worsen fatigue related decrement in performance including age, years of training/practice and clinical load prior to study participation.

ELIGIBILITY:
Inclusion Criteria:

* All attending anesthesiologists taking overnight call at Evanston Hospital will be eligible participants.

Exclusion Criteria:

* Resident physician or trainee, physician not taking overnight in house call.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical performance Score | 24 months
  Performance score on Stat c-section rating scale based on video rating by 2 raters

SECONDARY OUTCOMES:
Stanford Sleepiness Scale | 24months
  SSS scores in rested and fatigue arms

CONTACTS AND LOCATIONS:
Locations (1):
- Evanston Hospital, Evanston, Illinois, United States